CLINICAL TRIAL: NCT03268460
Title: Incidence of Renal Tubular Acidosis in Nephrology Unit in Assiut University Childern Hospital (AUCH)
Brief Title: Incidence of Renal Tubular Acidosis in Nephrology Unit in Assiut University Childern Hospital
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Sally Ezzat Shafik mikhail, principal investigator, Assiut University
Other Study IDs: RTA in childern
Record Dates: First submitted 2017-08-28; First posted 2017-08-31 (Actual); Last update posted 2017-09-01 (Actual); Status verified 2017-08

CONDITIONS: Renal Tubule Acidosis
MeSH Terms: conditions — Acidosis, Renal Tubular | interventions — Blood Gas Analysis; Acid-Base Equilibrium; Kidney Function Tests; Urinalysis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Arterial blood gases — blood PH, HCO3
Diagnostic Test: Blood anion gap — (Na+) - (Cl- + HCO3-)
Diagnostic Test: serum electrolytes — Na+ , K+ , Cl- and calcium
Diagnostic Test: renal function test — blood urea and serum creatinine
Diagnostic Test: urine analysis — urine PH, specific gravity, aminoaciduria, glycosuria, phospaturia and 24 hr urine calcium

SUMMARY:
Providing summarized information on the clinical and biochemical characteristics and types of renal tubular acidosis in children in Assiut University Childern Hospital.

DETAILED DESCRIPTION:
The term renal tubular acidosis (RTA) is applied to a group of transport defects in the reabsorption of bicarbonate (HCO3_), the excretion of hydrogen ion (H_), or both. This condition was first described in 1935, confirmed as a renal tubular disorder in 1946, and designated "renal tubular acidosis" in 1951. The RTA syndromes are characterized by a relatively normal GFR and a metabolic acidosis accompanied by hyperchloremia and a normal plasma anion gap.

RTA is classified into 4 major forms: distal, proximal, hyperkalemic and combined RTA. Distal RTA is associated with reduced urinary acid secretion, proximal RTA ( pRTA ) is characterized by impaired bicarbonate (HCO3_) reabsorption, hyperkalemic RTA is an acid-base disturbance generated by aldosterone deficiency or resistance and combined RTA is due to carbonic anhydrase II deficiency. Electrolyte and acid-base disturbances are key components of each disorder .

Patients with pRTA present with growth failure in the 1st yr of life. Additional symptoms can include polyuria, dehydration (from sodium loss), anorexia, vomiting, constipation, and hypotonia. Patients with primary Fanconi syndrome have additional symptoms, secondary to phosphate wasting, such as rickets. Hypokalemia and related symptoms are also restricted to cases with the Fanconi syndrome.

Distal RTA shares features with those of pRTA, including non-anion gap metabolic acidosis and growth failure; distinguishing features of distal RTA include nephrocalcinosis and hypercalciuria Combined proximal and distal RTA is a type observed as the result of inherited carbonic anhydrase II deficiency in different organs and systems.

Patients with type IV RTA can present with growth failure in the first few years of life. Polyuria and dehydration (from salt wasting) are common. Laboratory tests reveal a hyperkalemic non-anion gap metabolic acidosis. Urine may be alkaline or acidic. Elevated urinary sodium levels with inappropriately low urinary potassium levels reflect the absence of aldosterone effect .

The first step in the evaluation of a patient with suspected RTA is to confirm the presence of a normal anion gap metabolic acidosis, identify electrolyte abnormalities, assess renal function, and rule out other causes of bicarbonate loss such as diarrhea .

The mainstay of therapy in all forms of RTA is bicarbonate replacement. Patients with pRTA often require large quantities of bicarbonate, up to 20 mEq/kg/24 hr. The base requirement for distal RTAs is generally in the range of 2-4 mEq/kg/24 hr, although patients' requirements can vary. Patients with type IV RTA can require chronic treatment for hyperkalemia with sodium potassium exchange resin .

ELIGIBILITY:
Inclusion Criteria:

* Age : From 1 year to 18 year.
* Sex : Both sex male and female.
* All cases presented with hypokalemia and normal anion gap hyperchloremic metabolic acidosis with a relatively normal glomerular filteration rate.

Exclusion Criteria:

* Acute diarrhea .
* Urinary diversions.
* Post hypocapnia.
* Postobstructive diuresis.
* Interstitial nephritis.
* Active urinary tract infection.
* Intake of medications interfere with urinary acidification.

Ages: 1 Year to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: • All cases presented with hypokalemia and normal anion gap hyperchloremic metabolic acidosis with a relatively normal glomerular filteration rate.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2018-01 (Estimated); Primary Completion 2019-01 (Estimated); Study Completion 2019-01 (Estimated)

PRIMARY OUTCOMES:
percentage of cases with newly diagnosed renal tubular acidosis | Baseline
  percentage of cases presented by metabolic acidosis , failure to thrive and polyuria and diagnosed as RTA by arterial blood gases, blood anion gap, serum electrolytes, kidney function tests and urine analysis.

SECONDARY OUTCOMES:
percentage of cases with each type of RTA | Baseline
  this is by measurement of serum K+ and urine PH. normal or low level of serum K+ with urine PH < 5,5 with proximal RTA, while normal or low level of serum K+ with urine PH > 5,5 with distal RTA. high level of serum K+ with urine PH < 5,5 with hyperkalemic type 4 RTA, while high level of serum K+ with urine PH > 5,5 with voltage defect distal RTA